CLINICAL TRIAL: NCT01680549
Title: Pain Control With Total Knee Replacement: Does Gabapentin Affect Narcotic Usage and Functional Outcome? A Randomized Controlled Trial.
Brief Title: Pain Control With Total Knee Replacement
Acronym: L12-078
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L12-078
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin 600mg PO pre-operatively and continued postoperatively 300 mg PO q8 hours x 3 days.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo 600 mg po preoperatively and continued postoperatively 300 mg po q8hours X 3 days
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 600mg PO pre-operatively and continued postoperatively 300 mg PO q8 hours x 3 days.
  Other Names: Fanatrex; Gabarone; Gralise; Horizant; Neurontin

SUMMARY:
The purpose of this project is to study the effects of gabapentin on pain control in the perioperative and post-operative period of total knee arthroplasty.

DETAILED DESCRIPTION:
Being able to understand and better control pain in patients undergoing total knee arthroplasty will help in many different areas of medicine. Gabapentin is one pain control modality that has been used by many different orthopaedic surgeons with excellent retrospective results. Gabapentin, however, has never been studied, to the investigators knowledge, in a prospective randomized fashion in the United States for total knee arthroplasty. This study will be the first of its kind to truly compare the effects of gabapentin, a drug that has been proven safe in many other areas of medicine, with placebo for total knee arthroplasty by analyzing post-operative narcotic usage, function and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 25 years old

  * Primary osteoarthritis of the knee
  * Must be undergoing unilateral total knee arthroplasty
  * Anesthesia assesment score I, II, or III

Exclusion Criteria:

* Severe joint malalignment (defined as varus/valgus angle > 20 deg)

  * Use of gabapentin pre-operatively
  * History of chronic pain (currently under treatment)
  * History of substance abuse
  * Impaired kidney function (defined as creatinine > 1.5)
  * Epilepsy (currently on medication for treatment)
  * Known allergy to Gabapentin
  * Known history of depression or suicidal thoughts and behaviors
  * Anyone who is not a candidate for general anesthesia or any other portion of the investigator's standard of care.

Ages: 25 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W Brindley, MD, Principal Investigator — TTUHSC dept. Orthopaedic Surgery
Locations (1):
- TTUHSC Orthopaedic Surgery MS 9436, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo 1 tab PO preoperatively and 1 tab PO continued postoperatively q8hours X 3 days
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 25 | 25
Completed | 20 | 17
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (10.1) | 63.1 (11.2) | 62.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Patient Pain Scores
Description: Patient's pain assessed by the Visual Analog Scale (VAS - Units on a scale) on postoperative days 0, 1 and 2.
  Scale range: 0-100 Higher Values = More Pain
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: units on a scale- VAS
Groups:
- Placebo: Placebo- Comparator
- Gabapentin: Active pain medicine
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 17 | 20
units on a scale- VAS
  Day 0 | 33.6 (23.3) | 40.0 (26.1)
  Day 1 | 34.9 (26.6) | 46.3 (30.5)
  Day 2 | 38.0 (15.9) | 39.6 (18.8)

2. Secondary Outcome: Narcotics Consumption
Description: Narcotics consumption was recorded on postoperative days 0, 1, and 2.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Morphine dose equivalents
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 20 | 17
Morphine dose equivalents
  Day 0 | 4.16 (9.02) | 7.40 (9.10)
  Day 1 | 11.53 (13.90) | 25.02 (17.28)
  Day 2 | 11.61 (10.78) | 21.62 (17.28)

3. Secondary Outcome: Knee Range of Motion
Description: Patient knee range of motion was assessed on postoperative days 0, 1 and 2.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- Gabapentin: Active pain control Medicine
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 17 | 20
Degrees
  Day 0 | 53.12 (17.72) | 57.85 (17.70)
  Day 1 | 66.81 (20.54) | 62.74 (19.44)
  Day 2 | 67.47 (23.13) | 65.94 (15.20)

4. Secondary Outcome: Patient Restfulness
Description: Percentage of self reported patient restfulness was recorded on postoperative days 0, 1 and 2.
Time Frame: 3 days
Measure: Number; unit: Percent(%) of participants
Groups:
- Placebo: Placebo comparator
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 17 | 20
Percent(%) of participants
  Day 0 | 35.3 | 55.0
  Day 1 | 52.9 | 75.0
  Day 2 | 58.5 | 65.0

ADVERSE EVENTS:
Time Frame: AE data was collected through the completion of 2 weeks post op visit unless an AE to follow
Arm/Group | Placebo | Gabapentin
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Gabapentin (N=20)
Postoperative illeus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Traumatic foley insertion (Renal and urinary disorders) | 0 (0) | 1 (1)
Bradycardia and vasovagal syncope (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No